

| Official Title: A pilot mixed methods study of a camouflaged WeChat |
|-----------------------------------------------------------------------|
| mini-program-based intervention for women victims of intimate partner |
| violence |
| NCT number: Not yet assigned |
| Date of the document: 2024 12 20 |



### **Information Sheet**

# A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

You are invited to participate in a research study conducted by Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong.

# Purpose of the research

This study aims to determine the feasibility and acceptability of a camouflaged WeChat miniprogram-based WOMEN (abbreviated from Work Out for MEntal & Nutritional) Health intervention for women victims of intimate partner violence (IPV).

### **Procedures**

During the formative stage, key informants (ie., IPV experts, local non-governmental organization representatives, government officials, emergency physicians and nurses, community nurses, social workers, and police officers) will be invited to share practice and experience of working with women victims of IPV, beliefs about IPV and victims, availability of IPV resources, and opinions on the WeChat mini-program prototype. Key informant interviews will last approximately 30 minutes and be audio-recorded.

### **Risks**

The study is anticipated to have minimal risk as as time burden or discomfort due to IPV-related discussion.

# **Compensation and benefits for participation**

There are no direct financial benefits. You may gain informational benefits through participating in the study. For the society, results of this study can provide basis for future education, practice, and research to better respond to IPV.

## Confidentiality and data retention

All information will be kept strictly confidential. All data (e.g., recordings and transcripts) will be stored anonymously, and only the research team will have access to information recorded during the study. For audio recordings, your name will not be mentioned, and it will not be possible to identify your identity through your voice. Combination of English letters and numbers instead of real name will be used to represent individual participant. Your signed consent form will be stored separately from your personal information to further protect your privacy. All research data and personal information will be stored on an encrypted hard drive accessible only to the research team. You have the right to access personal data and publicly available study results if needed. All information can be retrieved or destroyed upon your request. All data will be destroyed 5 years after the completion of the research project.

By consenting to participate in this study, you expressly authorize:

• the principal investigator and his research team and the ethics committee (Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster) responsible for overseeing this study to get access to, to use, and to retain your



- personal data for the purposes and in the manner described in this informed consent process; and
- the relevant government agencies (e.g., the Hong Kong Department of Health) to get access to your personal data for the purposes of checking and verifying the integrity of study data and assessing compliance with the study protocol and relevant requirements.

# Participation and withdrawal

Your participation is voluntary. This means that you can choose to stop at any time without negative consequences.

## **Funding source**

This study is supported by the Health and Medical Research Fund (HMRF) of the Government of the Hong Kong Special Administrative Region. The funding source has no role in the study design, data collection, analysis, interpretation, or manuscript preparation.

# **Questions and concerns**

If you have any questions about the research, please feel free to contact Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong, by telephone (9544 9998) or email (qli1@hku.hk). This proposal has been reviewed and approved by the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster. If you have any questions regarding your rights as a research participant, please contact the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster by telephone (2255 4086) or email (hkwirb@ha.org.hk).



# A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

# **PARTICIPANT CONSENT FORM**

Participant ID:

Name of Researcher: Dr. Quanlei Li. Research Assistant Professor

| 1. | I confirm that I have read above study and have had | | |
|---|---|---|---|
| 2. | I understand that my par<br>withdraw at any time, wi<br>legal rights being affected | | |
| 3. | I agree to participate in th | | |
| Name of Subject | | Date Signat | ure |
| Nai | me of Investigator | Date Signat | ure |



### **Information Sheet**

# A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

You are invited to participate in a research study conducted by Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong.

### Purpose of the research

This study aims to determine the feasibility and acceptability of a camouflaged WeChat miniprogram-based WOMEN (abbreviated from Work Out for MEntal & Nutritional) Health intervention for women victims of intimate partner violence (IPV).

### **Procedures**

During the formative stage, women victims of IPV are invited for focus group interviews to share experiences and beliefs about IPV, awareness and utilization of IPV resources, and opinions on the WeChat mini-program prototype. Each focus group will have five participants, take place in a quiet and safe space. Focus group interviews will last approximately 60 min and be audio-recorded.

### **Risks**

The study is anticipated to have minimal risk as emotional distress and confidentiality breaches due to IPV-related intervention, discussion, and data collection.

#### **Compensation and benefits for participation**

There are no direct financial benefits. You may gain informational benefits through participating in the study. For the society, results of this study can provide basis for future education, practice, and research to better respond to IPV.

## **Confidentiality and data retention**

All information will be kept strictly confidential. All data (e.g., recordings and transcripts) will be stored anonymously, and only the research team will have access to information recorded during the study. For audio recordings, your name will not be mentioned, and it will not be possible to identify your identity through your voice. Combination of English letters and numbers instead of real name will be used to represent individual participant. Your signed consent form will be stored separately from your personal information to further protect your privacy. All research data and personal information will be stored on an encrypted hard drive accessible only to the research team. You have the right to access personal data and publicly available study results if needed. All information can be retrieved or destroyed upon your request. All data will be destroyed 5 years after the completion of the research project.

By consenting to participate in this study, you expressly authorize:

• the principal investigator and his research team and the ethics committee (Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster) responsible for overseeing this study to get access to, to use, and to retain your



- personal data for the purposes and in the manner described in this informed consent process; and
- the relevant government agencies (e.g., the Hong Kong Department of Health) to get access to your personal data for the purposes of checking and verifying the integrity of study data and assessing compliance with the study protocol and relevant requirements.

# Participation and withdrawal

Your participation is voluntary. This means that you can choose to stop at any time without negative consequences.

## **Funding source**

This study is supported by the Health and Medical Research Fund (HMRF) of the Government of the Hong Kong Special Administrative Region. The funding source has no role in the study design, data collection, analysis, interpretation, or manuscript preparation.

### **Questions and concerns**

If you have any questions about the research, please feel free to contact Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong, by telephone (9544 9998) or email (qli1@hku.hk). This proposal has been reviewed and approved by the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster. If you have any questions regarding your rights as a research participant, please contact the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster by telephone (2255 4086) or email (hkwirb@ha.org.hk).



Name of Investigator

# A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

# PARTICIPANT CONSENT FORM

Participant ID:

Name of Researcher: Dr. Quanlei Li, Research Assistant Professor

Please check box√

1. I confirm that I have read and understood the information sheet for the above study and have had the opportunity to ask questions. 

2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my care or legal rights being affected.

3. I agree to participate in the above study.

Signature

Date



## **Information Sheet**

# A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

You are invited to participate in a research study conducted by Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong.

## **Purpose of the research**

This study aims to determine the feasibility and acceptability of a camouflaged WeChat miniprogram-based WOMEN (abbreviated from Work Out for MEntal & Nutritional) Health intervention for women victims of intimate partner violence (IPV).

## **Procedures**

This study will invite 86 Chinese immigrant women who are screened positive for IPV by using the Chinese version of the Abuse Assessment Screen (AAS) from local community centers and women's shelters. If you decide to participate in this study, we will first ask you to complete an online questionnaire regarding your depressive symptoms, quality of life, IPV, and healthy behaviors. We will also measure your body weight and height to calculate the body mass index (BMI), defined as the ratio of body weight (kg) and height (m) squared. The process will take approximately 20 minutes to complete. You will then be randomly assigned to one of the following two groups:

- Group A: Participants will receive the WOMEN Health programme via a specifically developed WeChat mini-program, including disguised healthy lifestyle intervention, as well as genuine IPV intervention (empowerment and social support) accessed through the hidden user interfaces within the WeChat mini-program. Participants will receive a 60-min one-to-one interview as empowerment, and 12 weekly WeChat voice or telephone calls as social support.
- Group B: Participants will receive general knowledge on healthy lifestyle and 12 weekly calls about weight management and healthy lifestyle. After Group A complete the WOMEN Health programme, participants will also receive the same intervention delivered via the WeChat mini-program.

Each participant has a 50% chance of being assigned to either group. Both groups will receive a body scale free of charge for weight monitoring. Throughout the intervention, our research team will do our best to address any questions you may have about the process. At the end of the intervention, we will invite you to complete the online questionnaire again to assess changes in depressive symptoms, quality of life, IPV, BMI, and healthy behaviors. Additionally, after the intervention, we will invite about 12 participants from Group A to participate in an in-depth interview. You may be invited to share your experiences with the intervention, changes in IPV and lifestyle, and thoughts on usefulness and recommendations for the intervention. Interviews will last approximately 30 minutes and be audio-recorded.

#### Risks

The study is anticipated to have minimal risk as emotional distress and confidentiality breaches due to IPV-related intervention, discussion, and data collection.



## **Compensation and benefits for participation**

There are no direct financial benefits. A body weight scale will be provided as incentives for participation and used for body weight monitoring. You may gain empowerment and social support and informational benefits through participating in the study.

## Confidentiality and data retention

All information will be kept strictly confidential. Each questionnaire will be stored anonymously, and only the research team will have access to information recorded during the study. For audio recordings, your name will not be mentioned, and it will not be possible to identify your identity through your voice. Combination of English letters and numbers instead of real name will be used to represent individual participant. Your signed consent form will be stored separately from your personal information to further protect your privacy. All research data and personal information will be stored on an encrypted hard drive accessible only to the research team. You have the right to access personal data and publicly available study results if needed. All information can be retrieved or destroyed upon your request. All data will be destroyed 5 years after the completion of the research project.

By consenting to participate in this study, you expressly authorize:

- the principal investigator and his research team and the ethics committee (Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster) responsible for overseeing this study to get access to, to use, and to retain your personal data for the purposes and in the manner described in this informed consent process; and
- the relevant government agencies (e.g., the Hong Kong Department of Health) to get access to your personal data for the purposes of checking and verifying the integrity of study data and assessing compliance with the study protocol and relevant requirements.

## Participation and withdrawal

Your participation is voluntary. This means that you can choose to stop at any time without negative consequences.

## **Funding source**

This study is supported by the Health and Medical Research Fund (HMRF) of the Government of the Hong Kong Special Administrative Region. The funding source has no role in the study design, data collection, analysis, interpretation, or manuscript preparation.

#### **Questions and concerns**

If you have any questions about the research, please feel free to contact Dr. Quanlei Li, a Research Assistant Professor in the School of Nursing at the University of Hong Kong, by telephone (9544 9998) or email (qli1@hku.hk). This proposal has been reviewed and approved by the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster. If you have any questions regarding your rights as a research participant, please contact the Institutional Review Board of the University of Hong Kong/Hospital Authority Hong Kong West Cluster by telephone (2255 4086) or email (hkwirb@ha.org.hk).



**Participant ID:** 

A pilot mixed methods study of a camouflaged WeChat mini-program-based intervention for women victims of intimate partner violence

# PARTICIPANT CONSENT FORM

Name of Researcher: Dr. Quanlei Li, Research Assistant Professor

Please check box√

1. I confirm that I have read and understood the information sheet for the above study and have had the opportunity to ask questions. □

2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my care or legal rights being affected. □

3. I agree to participate in the above study, including the randomized controlled trial and, if invited, the post-intervention interview.

| Initial of Subject | Date | |
|----------------------|------|---------------|
| Name of Investigator | Date | <br>Signature |